CLINICAL TRIAL: NCT06765876
Title: Safety and Efficacy of Anti-CD123 Chimeric Antigen Receptor-Modified Autologous T Cells (CART123) in Patients With Relapsed/Refractory CD123+ Hematologic Malignancies: A Dose Escalation, Open-Label, Phase I Study
Brief Title: CART123 T Cells in Relapsed or Refractory CD123+ Hematologic Malignancies: A Dose Escalation Phase I Trial
Acronym: UHKT-CAR123-01
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Institute of Hematology and Blood Transfusion, Czech Republic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHKT-CAR123-01; 2022-503165-30-00 (EU CTIS Number)
Record Dates: First submitted 2024-12-18; First posted 2025-01-09 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-01

CONDITIONS: Leukemia, Myeloid, Acute(AML); Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes (MDS); Blastic Plasmacytoid Dendritic Cell Neoplasm (BPDCN)
Keywords: CAR123 T lymphocytes; CART123; CD123+ Hematologic Malignancies; Anti-CD123; Chimeric Antigen Receptor (CAR) T Cells; Autologous T Cells; Hematopoietic Malignancies; Immunotherapy; Personalized Medicine; Biological Therapy; Phase I Clinical Trial; Acute Lymphoblastic Leukemia, in Relapse; Acute Lymphoblastic Leukemia, Refractory; Relapsed Myelodysplastic syndrome; Relapsed Blastic Plasmacytoid Dendritic Cell Neoplasm; Acute Myeloid Leukaemia Recurrent
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes; Blastic Plasmacytoid Dendritic Cell Neoplasm; Hematologic Neoplasms

STUDY DESIGN:
Intervention Model Description: Experimental: Autologous CAR123 T lymphocytes
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): Experimental: Autologous CAR123 T lymphocytes
  Interventions: Biological: Autologous CAR123 T lymphocytes

INTERVENTIONS:
Biological: Autologous CAR123 T lymphocytes — Anti-CD123 Chimeric Antigen Receptor (CAR) T-Cells (CART123)
  Other Names: CART123; CAR123 T Cells; Autologous T-cell Therapy

SUMMARY:
Adult patients with refractory or relapsed CD123+ hematologic malignancies, including acute myeloid leukemia, myelodysplastic syndrome, acute lymphoblastic leukemia, or blastic plasmocytoid dentritic cell neoplasm will be recruited in the trial. CART123 cells will be manufatured from blood of each patient. During the production of CAR123 cells, patients may receive appropriate bridging therapy. After cells are produced, participants will undergo a single course of lymphodepleting chemotherapy and receive a single dose of CAR123 T cells. The trial will establish the recommended dose for further studies, either the Maximum Tolerated Dose (MTD) or Maximum Feasible Dose (MFD). Patients must be eligible for hematopoietic stem cell transplantation in order to participate in the trial.

DETAILED DESCRIPTION:
This is an open-label, single arm study on up to 18 adult subjects with refractory or relapsed CD123+ AML, MDS, ALL or BPDCN. Following lymphodepleting conditioning regimen, the subjects will receive a single dose of autologous CAR123 T lymphocytes supplied by the sponsor´s manufacturing facility.

CART123 dose will be increased in three predefined steps using the accelerated Bayesian optimal interval (BOIN) design in order to establish recommended CART123 dose for further study, which will be either Maximum Tolerated Dose (MTD) or Maximum Feasible Dose (MFD), whichever is reached first.

Alternative dosing schedule will be adopted in case of dose limitation due to insufficient CART123 expansion during IMP manufacture.

Due to concern for potentially prolonged or irreversible hematologic toxicity of CART123, all patients recruited in the study must be eligible for hematopoietic stem cell transplantation (HSCT) and have a donor of allogeneic hematopoietic stem cells identified and cleared by the transplant center. Decision to perform HSCT will be made on a case-by-case basis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with AML, MDS-IB2, BPDCN or ALL positive for CD123 antigen, who meet one of disease specific criteria below:

   a) Patients with AML will be eligible if they meet one of the following criteria:

   i) Patient with refractory AML defined as failure to achieve CR or CRi after at least 2 cycles of induction chemotherapy or 1 cycle of high dose salvage regimen or 4 cycles of venetoclax with azacytidine OR

   ii) Second or subsequent relapse of AML OR

   iii) Relapse after allogeneic HSCT.

   b) Patients with ALL will be eligible if they meet one of following criteria:

   i) disease refractory to or relapsed after CAR-19 cell therapy OR

   ii) CD19 negative relapse ineligible for treatment with TKI inhibitors and inotuzumab ozogamicin.

   c) Patients with BPDCN will be eligible if they meet following criteria:

   i) Refractory or relapsing after chemotherapy with or without allogeneic stem cell transplantation.

   d) Patients with MDS-IB2 will be eligible if they meet one of following criteria:

   i) Disease refractory to at least four cycles of azacytidine or progression on azacytidine-based therapy OR

   ii) Disease refractory to induction chemotherapy OR

   iii) Relapse after haematopoietic stem cell transplantation.
2. CD123 expression on malignant cells confirmed by flow cytometry or by immunohistochemistry.
3. Age between 18 and 70 years.
4. Patient has a suitable donor for allogeneic hematopoietic stem cell transplantation. Workup and clearance of the donor must be completed before IMP administration.
5. Patient able to understand and sign informed consent.
6. Women of child-bearing potential: negative pregnancy test at enrolment (PSV) and at Visit 1.
7. Patient for whom there are no standard-of-care treatments available or such treatment options have been exhausted.

Exclusion Criteria:

1. Known hypersensitivity to any component of the IMP.
2. Allogeneic HSCT within 3 months prior to IMP administration.
3. Severe, uncontrolled active infection.
4. Life expectancy < 8 weeks.
5. Respiratory insufficiency (need for oxygen therapy).
6. Significant liver impairment: bilirubin > 50 µmol/L, AST or ALT > 4 times normal upper limit.
7. Acute kidney injury with serum creatinine > 180 µmol/L, oliguria or need for acute dialysis.
8. Heart failure with LVEF < 50% by echocardiography.
9. Presence of active grade 3 - 4 acute GvHD or severe chronic GvHD.
10. Serious uncontrolled neurological comorbidity.
11. Vaccination with live virus vaccines in the 4 weeks before IMP administration and within 90 days after the IMP dose.
12. Women: pregnancy or breast-feeding.
13. Subjects of fertile age, unless permanent sexual abstinence is their lifestyle choice:

    1. female patients of childbearing potential not willing to use a highly effective method of contraception during the study,
    2. male patients whose sexual partner(s) are women of childbearing potential who are not willing to use a highly effective method of contraception during the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-10-23 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of autologous CART123 cells | 28 Days, Months 24
  Cumulative incidence of IMP-related adverse events (AEs) graded by ASTCT consensus grading criteria for Cytokine Release Syndrome (CRS) and Immune effector cell-associated neurotoxicity syndrome (ICANS) and by Common Terminology Criteria for Adverse Events (CTCAE) v 5.0 for other AEs
Rate of hematological recovery | 14 Days, 28 Days, 1Year, Months 12, Months 24
  Rate of hematological recovery, defined as absolute neutrophil count (ANC) > 1x 10^9/L and platelet count > 20x10^9/L without transfusion support. Hematological recovery before and after HSCT will be evaluated separately.
A dose of CART123 cells for further study | 14 Days, 28 Days, 1year, Months 12, Months 24
  Incidence of dose-limiting toxicities (DLTs) and other safety data after IMP administration.

SECONDARY OUTCOMES:
Morphologic Leukemia Free State (MLFS). | at day 14 and 28 after IMP administration.
  Efficacy of IMP administration in patients with refractory or relapsed AML, MDS, BPDCN and ALL evaluated by rate of morphologic leukemia-free state (MLFS).
Complete Remission (CR) rate | at 28 days and at any later point after IMP administration, before and after HSCT.
  Efficacy of IMP administration in patients with refractory or relapsed AML, MDS, BPDCN and ALL evaluated by Complete Remission (CR) rate.
Median Overall Survival and Overall Survival | at one year after IMP administration.
  Efficacy of IMP administration in patients with refractory or relapsed AML, MDS, BPDCN and ALL evaluated by overall survival (OS)
Feasibility and need for allogeneic hematopoietic cell transplantation after IMP administration | within 28 days of IMP administration
  Proportion of patients who did not recover blood counts within 28 days of IMP administration, proportion of patients who received allogeneic haematopoietic stem cell transplantation, and who engrafted after transplant.

OTHER OUTCOMES:
Determination of persistence and phenotype of CART123 cells in peripheral blood and bone marrow. | Days 1, 3, 5, 7, 14, 28, 49, 70, 100. Months 6, 12, 24.
  Number (absolute and percentage of T lymphocytes) of CART123 cells in peripheral blood and bone marrow.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Vydra, MD, PhD, Principal Investigator — Institute of Hematology and Blood Transfusion, Prague, Czech Republic; Petr Lesný, MD, PhD, Study Director — Institute of Hematology and Blood Transfusion, Prague, Czech Republic
Locations (1):
- Ustav hematologie a krevni transfuze / Institute of Hematology and Blood Transfusion, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Beckermann TM, Luo W, Wilson CM, Veach RA, Wilson MH. Cognate restriction of transposition by piggyBac-like proteins. Nucleic Acids Res. 2021 Aug 20;49(14):8135-8144. doi: 10.1093/nar/gkab578. PMID: 34232995; PMCID: PMC8373079. — https://pubmed.ncbi.nlm.nih.gov/34232995/
- See also: Bire S, Ley D, Casteret S, Mermod N, Bigot Y, Rouleux-Bonnin F. Optimization of the piggyBac transposon using mRNA and insulators: toward a more reliable gene delivery system. PLoS One. 2013 Dec 3;8(12):e82559. doi: 10.1371/journal.pone.0082559. PMID: 24 — https://pmc.ncbi.nlm.nih.gov/articles/PMC3849487
- See also: Bôle-Richard, E., Fredon, M., Biichlé, S. et al. CD28/4-1BB CD123 CAR T cells in blastic plasmacytoid dendritic cell neoplasm. Leukemia 34, 3228-3241 (2020). https://doi.org/10.1038/s41375-020-0777-1 — https://www.nature.com/articles/s41375-020-0777-1
- See also: Di Stasi A, Tey SK, Dotti G, Fujita Y, Kennedy-Nasser A, Martinez C, Straathof K, Liu E, Durett AG, Grilley B, Liu H, Cruz CR, Savoldo B, Gee AP, Schindler J, Krance RA, Heslop HE, Spencer DM, Rooney CM, Brenner MK. Inducible apoptosis as a safety switch — https://pmc.ncbi.nlm.nih.gov/articles/PMC3236370/
- See also: Gill S, Tasian SK, Ruella M, Shestova O, Li Y, Porter DL, Carroll M, Danet-Desnoyers G, Scholler J, Grupp SA, June CH, Kalos M. Preclinical targeting of human acute myeloid leukemia and myeloablation using chimeric antigen receptor-modified T cells. Bloo — https://pmc.ncbi.nlm.nih.gov/articles/PMC3983612/
- See also: Hamada M, Nishio N, Okuno Y, Suzuki S, Kawashima N, Muramatsu H, Tsubota S, Wilson MH, Morita D, Kataoka S, Ichikawa D, Murakami N, Taniguchi R, Suzuki K, Kojima D, Sekiya Y, Nishikawa E, Narita A, Hama A, Kojima S, Nakazawa Y, Takahashi Y. Integration M — https://pmc.ncbi.nlm.nih.gov/articles/PMC6116345/
- See also: Hofmann S, Schubert ML, Wang L, He B, Neuber B, Dreger P, Müller-Tidow C, Schmitt M. Chimeric Antigen Receptor (CAR) T Cell Therapy in Acute Myeloid Leukemia (AML). J Clin Med. 2019 Feb 6;8(2):200. doi: 10.3390/jcm8020200. PMID: 30736352; PMCID: PMC64068 — https://pmc.ncbi.nlm.nih.gov/articles/PMC6406805/
- See also: Kaštánková I, Štach M, Žižková H, Ptáčková P, Šmilauerová K, Mucha M, Šroller V, Otáhal P. Enzymatically produced piggyBac transposon vectors for efficient non-viral manufacturing of CD19-specific CAR T cells. Mol Ther Methods Clin Dev. 2021 Aug 26;23:11 — https://pmc.ncbi.nlm.nih.gov/articles/PMC8482285/
- See also: KRÖGER, Nicolaus; GRIBBEN, John; CHABANNON, Christian; YAKOUB-AGHA, Ibrahim a EINSELE, Hermann (ed.). The EBMT/EHA CAR-T Cell Handbook. Online. Cham: Springer, 2022. ISBN 978-3-030-94353-0 (eBook). https://doi.org/10.1007/978-3-030-94353-0. — https://link.springer.com/book/10.1007/978-3-030-94353-0
- See also: Li X, Burnight ER, Cooney AL, Malani N, Brady T, Sander JD, Staber J, Wheelan SJ, Joung JK, McCray PB Jr, Bushman FD, Sinn PL, Craig NL. piggyBac transposase tools for genome engineering. Proc Natl Acad Sci U S A. 2013 Jun 18;110(25):E2279-87. doi: 10.10 — https://pubmed.ncbi.nlm.nih.gov/23723351/
- See also: Maloney DG, Liles TM, Czerwinski DK, Waldichuk C, Rosenberg J, Grillo-Lopez A, Levy R. Phase I clinical trial using escalating single-dose infusion of chimeric anti-CD20 monoclonal antibody (IDEC-C2B8) in patients with recurrent B-cell lymphoma. Blood. 1 — https://pubmed.ncbi.nlm.nih.gov/7522629/
- See also: Mardiana S, Gill S. CAR T Cells for Acute Myeloid Leukemia: State of the Art and Future Directions. Front Oncol. 2020 May 6;10:697. doi: 10.3389/fonc.2020.00697. PMID: 32435621; PMCID: PMC7218049. — https://pmc.ncbi.nlm.nih.gov/articles/PMC7218049/
- See also: Micklethwaite KP, Gowrishankar K, Gloss BS, Li Z, Street JA, Moezzi L, Mach MA, Sutrave G, Clancy LE, Bishop DC, Louie RHY, Cai C, Foox J, MacKay M, Sedlazeck FJ, Blombery P, Mason CE, Luciani F, Gottlieb DJ, Blyth E. Investigation of product-derived lym — https://pmc.ncbi.nlm.nih.gov/articles/PMC8532197/
- See also: Mueller KT, Waldron E, Grupp SA, Levine JE, Laetsch TW, Pulsipher MA, Boyer MW, August KJ, Hamilton J, Awasthi R, Stein AM, Sickert D, Chakraborty A, Levine BL, June CH, Tomassian L, Shah SS, Leung M, Taran T, Wood PA, Maude SL. Clinical Pharmacology of — https://pmc.ncbi.nlm.nih.gov/articles/PMC7433345/
- See also: Prommersberger S, Reiser M, Beckmann J, Danhof S, Amberger M, Quade-Lyssy P, Einsele H, Hudecek M, Bonig H, Ivics Z. CARAMBA: a first-in-human clinical trial with SLAMF7 CAR-T cells prepared by virus-free Sleeping Beauty gene transfer to treat multiple m — https://pmc.ncbi.nlm.nih.gov/articles/PMC8455317/
- See also: Mardiros A, Dos Santos C, McDonald T, Brown CE, Wang X, Budde LE, Hoffman L, Aguilar B, Chang WC, Bretzlaff W, Chang B, Jonnalagadda M, Starr R, Ostberg JR, Jensen MC, Bhatia R, Forman SJ. T cells expressing CD123-specific chimeric antigen receptors exhi — https://pmc.ncbi.nlm.nih.gov/articles/PMC3814731/
- See also: Riberdy JM, Zhou S, Zheng F, Kim YI, Moore J, Vaidya A, Throm RE, Sykes A, Sahr N, Bonifant CL, Ryu B, Gottschalk S, Velasquez MP. The Art and Science of Selecting a CD123-Specific Chimeric Antigen Receptor for Clinical Testing. Mol Ther Methods Clin Dev — https://pmc.ncbi.nlm.nih.gov/articles/PMC7393323/
- See also: Ruella M, Barrett DM, Kenderian SS, Shestova O, Hofmann TJ, Perazzelli J, Klichinsky M, Aikawa V, Nazimuddin F, Kozlowski M, Scholler J, Lacey SF, Melenhorst JJ, Morrissette JJ, Christian DA, Hunter CA, Kalos M, Porter DL, June CH, Grupp SA, Gill S. Dual — https://pmc.ncbi.nlm.nih.gov/articles/PMC5096828/
- See also: Bire S, Ley D, Casteret S, Mermod N, Bigot Y, Rouleux-Bonnin F. Optimization of the piggyBac transposon using mRNA and insulators: toward a more reliable gene delivery system. PLoS One. 2013 Dec 3;8(12):e82559. doi: 10.1371/journal.pone.0082559. PMID: 24 — https://pubmed.ncbi.nlm.nih.gov/24312663/
- See also: Stevens BM, Zhang W, Pollyea DA, Winters A, Gutman J, Smith C, Budde E, Forman SJ, Jordan CT, Purev E. CD123 CAR T cells for the treatment of myelodysplastic syndrome. Exp Hematol. 2019 Jun;74:52-63.e3. doi: 10.1016/j.exphem.2019.05.002. Epub 2019 May 25 — https://pmc.ncbi.nlm.nih.gov/articles/PMC7184766/
- See also: Tashiro H, Sauer T, Shum T, Parikh K, Mamonkin M, Omer B, Rouce RH, Lulla P, Rooney CM, Gottschalk S, Brenner MK. Treatment of Acute Myeloid Leukemia with T Cells Expressing Chimeric Antigen Receptors Directed to C-type Lectin-like Molecule 1. Mol Ther. — https://pmc.ncbi.nlm.nih.gov/articles/PMC5589064/
- See also: Tasian SK, Kenderian SS, Shen F, Ruella M, Shestova O, Kozlowski M, Li Y, Schrank-Hacker A, Morrissette JJD, Carroll M, June CH, Grupp SA, Gill S. Optimized depletion of chimeric antigen receptor T cells in murine xenograft models of human acute myeloid — https://pmc.ncbi.nlm.nih.gov/articles/PMC5409446/
- See also: Tipanee J, VandenDriessche T, Chuah MK. Transposons: Moving Forward from Preclinical Studies to Clinical Trials. Hum Gene Ther. 2017 Nov;28(11):1087-1104. doi: 10.1089/hum.2017.128. Epub 2017 Aug 22. PMID: 28920716. — https://pubmed.ncbi.nlm.nih.gov/28920716/
- See also: Wang Y, Xu Y, Li S, Liu J, Xing Y, Xing H, Tian Z, Tang K, Rao Q, Wang M, Wang J. Targeting FLT3 in acute myeloid leukemia using ligand-based chimeric antigen receptor-engineered T cells. J Hematol Oncol. 2018 May 2;11(1):60. doi: 10.1186/s13045-018-0603 — https://pmc.ncbi.nlm.nih.gov/articles/PMC5930553/
- See also: Wermke M, Kraus S, Ehninger A, Bargou RC, Goebeler ME, Middeke JM, Kreissig C, von Bonin M, Koedam J, Pehl M, Bornhäuser M, Einsele H, Ehninger G, Cartellieri M. Proof of concept for a rapidly switchable universal CAR-T platform with UniCAR-T-CD123 in re — https://pmc.ncbi.nlm.nih.gov/articles/PMC8176767/
- See also: Bishop DC, Clancy LE, Simms R, Burgess J, Mathew G, Moezzi L, Street JA, Sutrave G, Atkins E, McGuire HM, Gloss BS, Lee K, Jiang W, Maddock K, McCaughan G, Avdic S, Antonenas V, O'Brien TA, Shaw PJ, Irving DO, Gottlieb DJ, Blyth E, Micklethwaite KP. Deve — https://pubmed.ncbi.nlm.nih.gov/34010392/
- See also: Tang TCY, Xu N, Nordon R, Haber M, Micklethwaite K, Dolnikov A. Donor T cells for CAR T cell therapy. Biomark Res. 2022 Apr 1;10(1):14. doi: 10.1186/s40364-022-00359-3. PMID: 35365224; PMCID: PMC8973942. — https://pmc.ncbi.nlm.nih.gov/articles/PMC8973942/
- See also: Yusa K, Zhou L, Li MA, Bradley A, Craig NL. A hyperactive piggyBac transposase for mammalian applications. Proc Natl Acad Sci U S A. 2011 Jan 25;108(4):1531-6. doi: 10.1073/pnas.1008322108. Epub 2011 Jan 4. PMID: 21205896; PMCID: PMC3029773. — https://pmc.ncbi.nlm.nih.gov/articles/PMC3029773/